CLINICAL TRIAL: NCT06985797
Title: Effects of Funfitness Program With Music Tempo on Perceived Exertion, Flexibility, Balance and Cognition in Gym Going Females
Brief Title: Funfitness Program With Music Tempo on Perceived Exertion, Flexibility, Balance and Cognition in Gym Going Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0452
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Funfitness program without music (Experimental): Group A will undergo FunFitness program without music (Control Group)
  Interventions: Other: Funfitness program with no music
- Funfitness Program with slow music (Experimental): Group B will undergo FunFitness program with slow music (Experimental Group)
  Interventions: Other: funfitness program with slow music
- Funfitness program with fast music (Experimental): Group C will undergo FunFitness program with fast music (Experimental Group)
  Interventions: Other: Funfitness program with fast music

INTERVENTIONS:
Other: Funfitness program with no music — Group A will undergo FunFitness program without music (Control Group)
  Arms: Funfitness program without music
Other: funfitness program with slow music — Group B will undergo FunFitness program with slow music (Experimental Group)
  Arms: Funfitness Program with slow music
Other: Funfitness program with fast music — Group C will undergo FunFitness program with fast music (Experimental Group)
  Arms: Funfitness program with fast music

SUMMARY:
The FunFitness Program was developed in collaboration with the American Physical Therapy Association and it includes measures of flexibility, strength, balance, and aerobic Olympics. The program is designed to be delivered by physical therapists, physical therapy assistants, and students of these respective disciplines. The participating Special Olympics athletes and their coaches and families are made aware of any physical limitations identified during the screen, and both educational and therapeutic interventions are provided. Athletes who are identified as having significant limitations may receive a referral for formal physical therapy services or physician visit if indicated. Regular exercise is essential for physical and cognitive health, particularly in females. The FunFitness program, a novel exercise approach that incorporates music tempo, has gained popularity among gym-goers. This study will investigate the effects of the FunFitness program with music tempo on perceived exertion, flexibility, balance, and cognition in gym-going females.

This study design will be Randomized clinical trial. Forty-five gym-going females aged 18-30 who are consistently going to gym from previous six months will randomly assigned to the FunFitness program with fast music tempo, slow music tempo and no music group. The FunFitness program with music tempo was conducted three times a week for 6 weeks. In this study researcher will use RPE and Feeling scale for perceived exertion .Sit and Reach Flexibility Test and V-Sit to measure flexibility.

DETAILED DESCRIPTION:
To determine the effects of funfitness program with music tempo on perceived exertion, flexibility, balance and cognition in gym going females.

ELIGIBILITY:
Inclusion Criteria:

Females Age between 18 to 30 years (12) Females who are going to the gym for the previous 6 months (13). Females having cognition value of more than 50

Exclusion Criteria:

Any kind of musculoskeletal injury (10) Any systematic illness : Hypertension or Diabetes Any trauma like fracture (14) Females with neurological problems (15)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Ratings of perceived exertion (RPE) scale | 6 weeks
  Illinois agility test is used to test running agility using various turns and movements Participants should lie on their front and hands by their shoulders. On the 'Go' command, the stopwatch is started, and the athlete gets up as quickly as possible and runs forwards ten meters to run around a cone, then back ten meters, then runs up and back through a slalom course of four cones. Finally, the athlete runs another ten meters up and back past the finishing cone, at which the timing is stopped. the point that best represents how hard you are working. The validity of RPE scale is 0.607. The reliability of this scale is 0.86.
Feeling scale | 6 weeks
  While participating in exercise it is quite common to experience changes in mood.. A scale has been designed to measure such responses [experimenter presents scale]. This scale is presented as an 10 points bipolar good/bad format. At five-minute intervals you are required to select the figure that best represents your feelings . I will tell you when you need to respond to this scale
V SIT | 6 weeks
  The Vsit test is used to measure flexibility. In this test, the participant will sit on floorwith leg straight. Then the participant will lean forward and reach towards toes, keeping knees straight. Hold this position for 1-2 seconds. Return to starting position.
Sit-and-reach flexibility test | 6 weeks
  The sit-and-reach test measures the flexibility of the lower back and hamstrings. In the past, there has not been consensus with regard to the validity and reliability of the test. Nevertheless, recent studies suggest that the criterion-related validity of the sit-and-reach test is moderate whereas the reliability is suggested to be acceptable. In the present study, the sit- and-reach test was performed using the procedures outlined in the ACSM manual. (14) .The reliability of this test is 0.89-0.98.The validity of this test is 0.46-0.67.
STAR EXCURSION BALANCE TEST | 6 weeks
  Dynamic standing balance will be assessed using the SEBT. Participants will be asked to stand on single leg in the center of star shaped figure on the floor. Then reach for points on the star with opposite leg, keeping the standing leg straight. Touch the point and return to the starting position. Repeat for all points on the star. Perform on both legs.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Punjab Squash Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang ZX, Su R, Li H, Dang P, Zeng TA, Chen DM, Wu JG, Zhang DL, Ma HL. Changes in Hippocampus and Amygdala Volume with Hypoxic Stress Related to Cardiorespiratory Fitness under a High-Altitude Environment. Brain Sci. 2022 Mar 8;12(3):359. doi: 10.3390/brainsci12030359. PMID 35326315
- [Background] Niedermeier M, Weiss EM, Steidl-Muller L, Burtscher M, Kopp M. Acute Effects of a Short Bout of Physical Activity on Cognitive Function in Sport Students. Int J Environ Res Public Health. 2020 May 23;17(10):3678. doi: 10.3390/ijerph17103678. PMID 32456170
- [Background] Barranco-Ruiz Y, Villa-Gonzalez E. Health-Related Physical Fitness Benefits in Sedentary Women Employees after an Exercise Intervention with Zumba Fitness(R). Int J Environ Res Public Health. 2020 Apr 11;17(8):2632. doi: 10.3390/ijerph17082632. PMID 32290490
- [Background] Lin HM, Kuo SH, Mai TP. Slower tempo makes worse performance? The effect of musical tempo on cognitive processing speed. Front Psychol. 2023 Feb 24;14:998460. doi: 10.3389/fpsyg.2023.998460. eCollection 2023. PMID 36910785
- [Background] Barene S, Holtermann A, Oseland H, Brekke OL, Krustrup P. Effects on muscle strength, maximal jump height, flexibility and postural sway after soccer and Zumba exercise among female hospital employees: a 9-month randomised controlled trial. J Sports Sci. 2016 Oct;34(19):1849-58. doi: 10.1080/02640414.2016.1140906. Epub 2016 Feb 5. PMID 26849477
- [Background] Norouzi E, Hosseini F, Vaezmosavi M, Gerber M, Puhse U, Brand S. Zumba dancing and aerobic exercise can improve working memory, motor function, and depressive symptoms in female patients with Fibromyalgia. Eur J Sport Sci. 2020 Aug;20(7):981-991. doi: 10.1080/17461391.2019.1683610. Epub 2019 Nov 7. PMID 31630663
- [Background] Edworthy J, Waring H. The effects of music tempo and loudness level on treadmill exercise. Ergonomics. 2006 Dec 15;49(15):1597-610. doi: 10.1080/00140130600899104. PMID 17090506
- [Background] Donath L, Roth R, Hohn Y, Zahner L, Faude O. The effects of Zumba training on cardiovascular and neuromuscular function in female college students. Eur J Sport Sci. 2014;14(6):569-77. doi: 10.1080/17461391.2013.866168. Epub 2013 Dec 10. PMID 24320999
- [Background] Chalhoub NE, Luggen ME. Screening for cognitive dysfunction in systemic lupus erythematosus: the Montreal Cognitive Assessment Questionnaire and the Informant Questionnaire on Cognitive Decline in the Elderly. Lupus. 2019 Jan;28(1):51-58. doi: 10.1177/0961203318815299. Epub 2018 Nov 27. PMID 30482092